CLINICAL TRIAL: NCT04867057
Title: A Phase 1 FIH, Randomized, Double Blind, Placebo Controlled, SAD/MAD Study to Assess Safety, Tolerability, PK/PD and Food Effect of Trichomylin in Healthy Adult Participants and Preliminary Efficacy in Management of Chronic OA Pain
Brief Title: Trichomylin® Safety, Tolerability & Pharmacokinetics in Healthy Adults and First in Human Osteoarthritis Pain Evaluation
Acronym: HOPE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ZYUS Life Sciences Inc. (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry); ZYUS Life Sciences Australia Pty Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Z-TRI-10001
Record Dates: First submitted 2021-04-16; First posted 2021-04-30 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Healthy; Osteoarthritis
Keywords: Cannabinoid; Safety and Tolerability; Pharmacokinetics; Pharmacodynamics; Chronic Pain
MeSH Terms: conditions — Osteoarthritis; Chronic Pain | interventions — Sagittal Abdominal Diameter; mycophenolic adenine dinucleotide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental: Trichomylin for SAD (Experimental): 18 out of 24 subjects were randomized to receive Trichomylin in a single dose.
  Interventions: Drug: Trichomylin for SAD
- Placebo Comparator: Placebo for SAD (Placebo Comparator): 6 out of 24 subjects were randomized to receive placebo in a single dose.
  Interventions: Drug: Placebo for SAD
- Experimental: Trichomylin for MAD (Experimental): 13 out of 17 subjects were randomized to receive Trichomylin in multiple doses.
  Interventions: Drug: Trichomylin for MAD
- Placebo Comparator: Placebo for MAD (Placebo Comparator): 4 out of 17 subjects were randomized to receive Placebo in multiple doses.
  Interventions: Drug: Placebo for MAD

INTERVENTIONS:
Drug: Trichomylin for SAD — Healthy subjects meeting eligibility criteria were randomized to each dose cohort (up to four dose ascending cohorts) to receive either Trichomylin or Placebo. The study drug (Trichomylin or Placebo) will be administered orally as a single dose.
  Arms: Experimental: Trichomylin for SAD
Drug: Placebo for SAD — Healthy subjects meeting eligibility criteria were randomized to each dose cohort (up to four dose ascending cohorts) to receive either Trichomylin or Placebo. The study drug (Trichomylin or Placebo) will be administered orally as a single dose.
  Arms: Placebo Comparator: Placebo for SAD
Drug: Trichomylin for MAD — Healthy subjects meeting eligibility criteria were randomized to each dose cohort (up to three cohorts) to receive either Trichomylin or Placebo. The study drug (Trichomylin or Placebo) will be administered daily oral doses for a total of 9 days.
  Arms: Experimental: Trichomylin for MAD
Drug: Placebo for MAD — Healthy subjects meeting eligibility criteria were randomized to each dose cohort (up to three cohorts) to receive either Trichomylin or Placebo. The study drug (Trichomylin or Placebo) will be administered daily oral doses for a total of 9 days.
  Arms: Placebo Comparator: Placebo for MAD

SUMMARY:
This is a first in human, randomized, double-blind, placebo-controlled SAD (with food effect) followed by a MAD study of Trichomylin® conducted in healthy adult participants.

DETAILED DESCRIPTION:
The study is designed to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and food effect of Trichomylin® in healthy adult participants.

A total of up to 40 participants were planned to be enrolled into Part A and Part B of the study. Part A consisted of 3 SAD cohorts (n = 8 per cohort) and Part B consisted of 2 MAD cohorts (n = 8 per cohort). Participants underwent a Screening period beginning up to 21 days for the SAD cohorts and 28 days for the MAD cohorts prior to randomization/dose administration. The Screening period was followed by admission to the clinical research unit (CRU), pre-dose assessment, post-dose assessment(s), and a final end of study (EOS)/follow-up visit.

Safety and tolerability endpoints are to report the percentage and severity of unexpected or serious adverse events, including clinically significant vital signs, laboratory test results, physical examination, and/or reported clinical symptoms, and use of concomitant medications. Other endpoints to be assessed are neurocognitive impairment, altered state of consciousness, and overall well-being.

Other assessments include pharmacokinetic (fasted and fed states) and pharmacodynamic endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female volunteers, aged 18 to 65 years (inclusive at the time of consent);
2. Must have a Body Mass Index (BMI) ≥ 18 to ≤ 32 kg/m2 with weight ≥ 50 kg at Screening;
3. Must have a negative urine drug screen at the Screening visit and the day before dosing (Day -1); one repeat urine drug may be conducted for a suspected false positive result;
4. Must be willing to abstain from the use of cannabis and other cannabinoid compounds (other than the study drug) for the duration of the study (from the time of Screening until the EOS visit);
5. Must be willing to abstain from smoking (including the use of tobacco or nicotine products and e-cigarettes) for the duration of the study (from the time of Screening until the EOS visit);
6. Must not have any hepatic and/or renal impairment as judged by the PI;
7. Must be willing and able to comply with all study procedures and be available for the duration of the study (from the time of Screening until the EOS visit);
8. Must not be currently using anti-depressants (selective serotonin reuptake inhibitors [SSRIs], monoamine oxidase inhibitors [MOAIs], serotonin-norepinephrine reuptake inhibitors [SNRIs], or tricyclic anti-depressants [TCAs]) for 14 days or 5 half-lives of the drug, whichever is longer, prior to IP administration, and for the duration of the study;
9. Must not have any current or past allergic or adverse reaction or known sensitivity to olive oil, gelatin, glycerin and titanium dioxide, or to cannabinoid-like substances (including but not limited to Dronabinol/Marinol/Nabilone/marijuana/cannabis/tetrahydrocannabinol [THC], cannabinoid oil);
10. Females must be non-pregnant and non-lactating and must use two forms ("double contraception") of acceptable, highly effective contraception from Screening and for 12 weeks following the last dose of study drug. Double contraception is defined as a condom AND one other form of the following:

    1. Established hormonal contraception (with an approved oral contraceptive pill [OCP]);
    2. Depot or injectable birth control;
    3. A vaginal ring or an intrauterine device ([IUD], with or without hormones); OR
    4. Documented evidence of surgical sterilization as a single form of birth control, at least 6 months prior to Screening (e.g., tubal ligation, hysterectomy, bilateral salpingectomy, or bilateral oophorectomy for women, OR vasectomy for men [with documented azoospermia 90 days after procedure] provided that partner is the sole sexual partner).

    Women not of childbearing potential must be post-menopausal (defined as cessation or regular menstrual periods for at least 12 months). Post-menopausal status will be confirmed through testing of follicle-stimulating hormone (FSH) consistent with post-menopausal state based on lab reference ranges.

    True subject abstinence for the duration of the study and 12 weeks after IP dosing is acceptable only when the subject has not been sexually active at all during their lifetime.

    Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhoea methods are not considered "true" abstinence and are not acceptable methods of contraception.

    Female participants who are in a long-term, same-sex, monogomous relationship are not required to use contraception.
11. Male subjects of childbearing potential will be required to use condoms from Screening until 12 weeks following the last dose of the study drug and to refrain from sperm donation during the same period. Male subjects not of childbearing potential are permanently sterile by bilateral orchidectomy or vasectomy (with documented azoospermia 90 days after procedure).

    Male participants who are in a long-term, same-sex, monogamous relationship are not required to use contraception.

    Male subjects should be informed that if a female partner becomes pregnant while he is enrolled in the study, contact with the female partner will be attempted to request her consent to collect pregnancy outcome information.
12. Women of childbearing potential must have a negative pregnancy test at Screening and Day -1 and be willing to have additional pregnancy tests, as required, throughout the study, at the Investigator's discretion;
13. Males must not donate sperm and females must not donate ova from Screening until 12 weeks after the last dose of the study drug.
14. Must agree to adhere to the current state and national advice regarding minimizing exposure to corona virus disease of 2019 (COVID-19) from the first Screening visit until the EOS visit;
15. Must be willing and able to provide written informed consent after the nature of the study has been explained and prior to the commencement of any study procedures;
16. Must be in good physical and mental health as determined by absence of any clinically significant (in the opinion of the Investigator) abnormalities based on medical history, physical examination, vital signs, triplicate 12-lead electrocardiogram (ECG), clinical laboratory evaluations, at Screening and prior to administration of the initial dose of study drug;
17. Must be able and willing to comply with all study requirements including:

    1. Confinement to the CRU prior to and during study drug administration and required follow-up periods for Part A SAD and Part B MAD
    2. Refraining from using the following:

    i. Any previous/current cannabis products within 2 months prior to Screening and throughout the duration of the study (from the time of Screening until the EOS visit); ii. Cannabis products (in the form of oil, vaporizer, or smoke) for the duration of the study; iii. Prescription medications 14 days prior to administration of the first dose of study drug; iv. Alcohol 48 hours prior to admission, and while confined to the CRU. In addition, participants must agree to refrain from regular use of alcohol (i.e. ˃ 10 units per week or ˃ 4 units on any given day for men and women [1 unit = 150mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]) for the duration of the study; v. Recreational drugs for the duration of the study.
18. For Part A SAD, participants must not have used cannabis or cannabinoid products within 2 months prior to Screening.

Exclusion Criteria:

1. Pregnant or lactating at Screening or planning to become pregnant (self or partner) at any time during the study and for 12 weeks after final study drug administration;
2. Has a past or present clinically significant condition, which would prevent or limit study assessments in accordance with the protocol, with particular reference to renal and/or hepatic impairment, OR it would be in the best interests of the participant to not participate;
3. Has been diagnosed with the following within 10 years of Screening: psychosis (secondary to, for example, substance abuse, major depression, a mood disorder with postpartum onset, bipolar disorder, schizophrenia, or borderline personality disorder), somatoform disorder(s) or chronic fatigue syndrome;
4. Has a current/active diagnosis of generalized anxiety disorder, panic disorder, obsessive compulsive disorder, post- traumatic stress disorder, a simple phobia(s), anorexia nervosa or bulimia nervosa;
5. Cognitive impairment and/or a psychiatric illness (e.g., dementia, Alzheimer's disease or psychosis), which in the opinion of the Investigator will prevent participants from reliably providing primary outcome data;
6. Has significant suicidal ideation as defined by the Columbia-Suicide Severity Rating Scale (C-SSRS) and Patient Health Questionnaire (PHQ-9);
7. History of abuse of substances such as opiates, amphetamines, barbiturates, cocaine, cannabis, hallucinogens within 12 months prior to Screening or positive urine drug screen at Screening or Day -1. A urine drug screen deemed positive due to prescription medications or for benzodiazepines or opioids is acceptable and inclusion is at the discretion of the Investigator;
8. Regular use of alcohol within one month prior to the Screening visit (i.e. more than 10 units of alcohol per week or 4 units on any given day [1 unit = 150mL of wine, 260 mL of beer, or 45mL of 40% alcohol]);
9. Symptomatic heart failure (per New York Heart Association [NYHA] guidelines), unstable angina, myocardial infarction, transient ischemic attack (TIA) or cerebrovascular accident (CVA) within 6 months prior to Screening;
10. Has an abnormal ECG of clinical relevance at Screening or Baseline, including but not limited to the following:

    1. QTcF interval > 450 msec
    2. Evidence of 2nd and 3rd degree atrioventricular (AV) block, or 1st degree AV block with PR interval > 200ms, left bundle branch block (LBBB) or right bundle branch block (RBBB) at Screening or Baseline. Incomplete RBBB will not permitted.
    3. Has a history of risk factors including hypokalemia, family history of Long QT Syndrome, or prior use of medications that prolong the QT/QTc interval
11. Has a resting heart rate < 45 beats/minute, > 100 beats/min upon one repeated measurement within 5 minutes;
12. Has abnormal blood pressure outside specified limits (90 mm Hg > Systolic > 140 mm Hg and/or 50 mm Hg > Diastolic > 90 mm Hg) upon repeated measurement;
13. Has clinically significant abnormalities in any of the clinical laboratory evaluations at Screening or Day -1 as determined by the Investigator;
14. Has a history of malignancy within the last 2 years except for adequately treated basal cell carcinoma, squamous cell skin cancer, superficial bladder tumors, or in situ cervical cancer. Participants with other curatively treated malignancies who have no evidence of metastatic disease and more than a 2-year disease-free interval may be entered following approval by the Study Medical Monitor (MM);
15. Has a history of major surgery within 6 months of Screening, OR has a history of minor surgery within the past month which would preclude inclusion as judged by the Investigator OR will not have fully recovered from surgery, OR has planned a surgery during the study;
16. Has current or past allergic or adverse reaction or known sensitivity to olive oil, gelatin, glycerin and titanium dioxide, or to cannabinoid-like substances (Dronabinol/Marinol/Nabilone/marijuana/cannabis/tetrahydrocannabinol [THC], cannabinoid oil);
17. Has known human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) infection, or tests positive for any of these viruses at Screening;
18. Use of the following in the 14 days prior to study drug administration or 5 half-lives, whichever is longer:

    1. Sedative medications (e.g., barbiturates and other central nervous system [CNS] depressants)
    2. Warfarin (Coumadin)
    3. Antipyrine
    4. Disulfiram (Antabuse)
    5. CYP3A4 inhibitors, inducers or substrates
    6. CYP2C9 inhibitors, inducers or substrates
    7. CYP2C19 inducers or substrates
    8. CYP2B6 substrates
    9. CYP1A2 substrates
    10. P-glycoprotein substrates

    Note: this includes grapefruit juice or related products, Sevilla orange juice or related products, and St John's wort.
19. Unable to swallow an oral tablet/capsule (medication) or consume up to 300 mL of water within 30 minutes;
20. Use of any IP or investigational medical device within 30 days prior to Screening, or 5 half-lives of the product (whichever is the longest), or current participation in an investigational study, or participation in more than 4 investigational drug studies within 1 year prior to Screening.
21. Refusal to maintain contraceptive practices (as defined by guidance) during the study and for 12 weeks after final study drug administration and for women of childbearing potential refusal to be screened for pregnancy for the duration of the study.
22. Study personnel as an immediate family or household member.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Percentage and severity of unexpected Serious Adverse Events (SAEs) | Through study completion, an average of 1 year
  To investigate the safety and tolerability of Trichomylin by assessment of the percentage and severity of SAEs following administration of oral soft-gel capsules in Single Ascending Dose (SAD Cohort) and Multiple Ascending Doses (MAD Cohort)

SECONDARY OUTCOMES:
Rate and extent of absorption of Trichomylin by assessment of the observed Maximum Plasma Concentration (Cmax) | SAD cohort: Day 1 through Day 21; MAD cohort: Day 1 through 30
  To assess the observed Maximum Plasma Concentration (Cmax) for SAD and MAD cohorts
Rate and extent of absorption of Trichomylin by assessment of the observed Time to Maximum Plasma Concentration (Tmax) | SAD cohort: Day 1 through Day 21; MAD cohort: Day 1 through 30
  To assess the observed Time to Maximum Plasma Concentration (Tmax) for SAD and MAD cohorts
Rate and extent of elimination of Trichomylin by assessment of the observed Apparent Terminal Elimination Rate Constant (Kel) | SAD cohort: Day 1 through Day 21; MAD cohort: Day 1 through 30
  To assess the observed Apparent Terminal Elimination Rate Constant (Kel) for SAD and MAD cohorts
Exposure of Trichomylin by assessment of area under the drug concentration-time curve (AUC). | SAD cohort: Day 1 through Day 21; MAD cohort: Day 1 through 30
  To assess the observed plasma exposure of Trichomylin AUC for SAD and MAD cohorts.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Wabnitz, Dr, Principal Investigator — CMAX clinical research
Locations (1):
- CMAX Clinical Research, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No